CLINICAL TRIAL: NCT06867536
Title: A Prospective, Single Arm, Phase Ⅱ Study to Evaluate the Efficacy and Safety of Hypofractionation Radiotherapy in Combination with Glofitamab in Relapsed/refractory Diffuse B-cell Lymphoma with Baseline High Tumor Burden
Brief Title: Hypofractionation Radiotherapy in Combination with Glofitamab in Relapsed/refractory Diffuse B-cell Lymphoma with Baseline High Tumor Burden
Acronym: GLOHRT-01
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Liling Zhang (Other)
Responsible Party: Sponsor-Investigator, Liling Zhang, chief physician, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHCT241108
Record Dates: First submitted 2025-02-11; First posted 2025-03-10 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Relapsed/Refractory Diffuse Large B-Cell Lymphoma (DLBCL); Lymphoma
Keywords: DLBCL; Glofitamab; radiotherapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma | interventions — glofitamab; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Glofitamab (Experimental): Utilizing intensity-modulated radiation therapy (IMRT); the radiation field follows the principles of involved site radiation therapy (ISRT). Total RT dose is 30 Gy/6 fraction, once daily, starting 8 days before Obinutuzumab pretreatment.
  An initial 1000 mg dose of Obinutuzumab will be administered as pretreatment 7 days prior to the first Glofitamab step-up dose Glofitamab is administered intravenously as step-up doses on day 8 (2.5 mg) and day 15 (10 mg) of cycle 1, followed by a dose of 30 mg on day 1 of cycles 2 through 8, maximum of 12 cycles (Q3W). The efficacy is evaluated after 2 cycles of Glofitamab. Those with disease progression will be withdrawn from the study. The remaining patients continue with an additional two cycles of Glofitamab (4 cycles in total) and then perform efficacy assessment. If the patients achieve a CR or PR, they will continue to complete the remaining treatment as planned.
  Interventions: Drug: Glofitamab + Obinutuzumab

INTERVENTIONS:
Drug: Glofitamab + Obinutuzumab — Obinutuzumab An initial 1000 mg dose of obinutuzumab will be administered as pretreatment 7 days prior to the first glofitamab step-up dose
  Glofitamab:
  Glofitamab was administered intravenously as step-up doses on day 8 (2.5 mg) and day 15 (10 mg) of cycle 1, followed by a dose of 30 mg on day 1 of cycles 2 through 8, maximum of 12 cycles (Q3W). The efficacy is evaluated after 2 cycles of glofitamab. Those with disease progression will be withdrawn from the study. The remaining patients continue with an additional two cycles of glofitamab (4 cycles in total) and then perform efficacy assessment. If the patients achieve a CR or PR, they will continue to complete the remaining treatment as planned. Patients are recommended to treat for 12 cycles (at least 8 cycles, depending on tumor regression in patients) or until disease progression or unacceptable toxicity, whichever occurs first

SUMMARY:
Glofitamab has shown efficacy and safety in the treatment of patients with relapsed/refractory diffuse large B-cell lymphoma (R/R DLBCL) and has been approved for marketing in China. However, in patients with baseline high tumor burden, the complete response (CR) rate is relatively lower compared with patients without. There is still a need to improve the efficacy of glofitamab in patients with high tumor burden. Previous studies have shown that hypofractionation radiotherapy (HRT) may induce T cell immune responses and improve the tumor microenvironment . Evidence shows that radiotherapy (RT) improves chimeric antigen receptor T-cell (CAR-T) efficacy as a bridging therapy . Based on the experience of RT combined with CAR-T, bispecific antibodies, as another T-cell therapy, may also demonstrate synergistic effects when combined with HRT, especially in those patients with bulky disease. This study will enroll R/R DLBCL patients with high tumor burden to assess the efficacy and safety of glofitamab in combination with HRT and to explore a new treatment model for R/R DLBCL patients with high tumor burden at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Aged 18-75 years at the time of signing the informed consent, willing to follow and able to complete all study procedures.
* Expected survival ≥ 12 weeks.
* ECOG performance status score of 0-2 points ;
* Patients with CD20-positive DLBCL confirmed by pathological histology; (unspecified DLBCL, HGBCL, PMBCL, FL-transformed DLBCL).
* R/R DLBCL who have received at least one line of systemic treatment (including at least 2 cycles of rituximab-containing immunochemotherapy).
* Baseline high tumor burden, defined as tumor diameter > 6 cm and/or TMTV > 128.7 mL .
* HIV test results were negative at screening, except for the following: HIV-positive patients who have been receiving stable antiretroviral therapy and CD4 count ≥ 200/µL before enrollment Patients with undetectable viral load can be enrolled.
* Women of childbearing age with negative urine or blood pregnancy test within 7 days before enrollment need to agree to take effective contraceptive measures during treatment and follow-up.

Exclusion Criteria:

* Individuals who have drug allergies or metabolic disorders to the drugs in this protocol.
* Previous recipients of allogeneic organ transplants.
* Individuals who received systemic immunotherapy within 4 weeks or 5 half-lives (whichever is shorter) of the drug.
* Anti-cancer drug treatment within 28 days before the start of treatment
* Prior radiotherapy in the mediastinum/pericardium area; radiation therapy for non-target lesion sites is allowed.
* History of severe or extensive cardiovascular disease.
* Recent major surgery (within 4 weeks before the start of Cycle 1), excluding diagnostic surgeries.
* Currently suffering from active CNS lymphoma.
* Known or suspected history of hemophagocytic lymphohistiocytosis (HLH)
* Current or previous history of concurrent Waldenström's macroglobulinemia.
* Known active infection at the time of enrollment in the study.
* Immune-related adverse events that appeared during prior immunotherapy: ≥Grade 3 adverse events, except for Grade 3 endocrine diseases controlled by alternative therapies. Grade 1 or 2 adverse events that did not return to baseline levels after stopping treatment.
* History of autoimmune diseases (long-standing or well-controlled autoimmune diseases, hypothyroidism, immune thrombocytopenic purpura, and well-controlled Type I diabetes are excluded).
* Abnormal coagulation function: INR or PT >1.5× upper limit of normal (ULN), PTT or aPTT >1.5× ULN.
* Suspected or latent tuberculosis (confirmed by positive IFNγ release test)
* Active hepatitis B virus (HBV) infection/positive HCV RNA test for hepatitis C virus (HCV)/HIV seropositive.
* Previously suffered from other invasive malignancies, excluding early-stage cervical cancer, basal cell carcinoma of the skin, and thyroid cancer .
* Pregnant or breastfeeding, or planning to become pregnant during the study period or within 18 months after pre-treatment with obinutuzumab or within 2 months after the last dose of glofitamab (whichever is longer).
* Other concurrent uncontrolled medical conditions that, in the investigator's opinion, would affect the patient's participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | From enrollment to the end of treatment at 8 cycles (each cycle is 21 days)
  defined as the percentage of patients whose best overall response was a CR according to the 2014 Lugano Response Criteria (Cheson, et al. 2014); as determined by the investigator

SECONDARY OUTCOMES:
Best response rate | From enrollment to the end of treatment at 8 cycles (each cycle is 21 days)
  defined as the proportion of patients whose best overall response is a PR or CR using 2014 Lugano Response Criteria (Cheson, et al. 2014)
DoCR | from the initial occurrence of a documented CR until documented disease progression or death due to any cause, assessed up to 48 months
  defined as the time from the initial occurrence of a documented CR until documented disease progression or death due to any cause, whichever occurs first,. This will be evaluated using investigator assessment based on the 2014 Lugano Classification (Cheson, et al. 2014).
PFS | the time from the first study treatment to the first occurrence of disease progression or death from any cause, whichever occurs first, assessed up to 48 months
  defined as the time from the first study treatment to the first occurrence of disease progression or death from any cause, whichever occurs first. PFS will be assessed by the investigator, using the 2014 Lugano classification (Cheson et al. 2014
OS | the time from the first study treatment to the date of death from any cause, assessed up to 48 months
  defined as the time from the first study treatment to the date of death from any cause.

IPD SHARING:
Plan to Share IPD: No